CLINICAL TRIAL: NCT00003824
Title: The Effect of Fluoroquinolones on the Disease-Free Interval in Patients With Stage Ta Transitional Cell Carcinoma of the Bladder
Brief Title: S9809, Ciprofloxacin Compared With Cephalexin in Treating Patients With Bladder Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Permanently Closed Due to Poor Accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066978; S9809 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2004-04-14 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Bladder Cancer
Keywords: stage 0 bladder cancer; recurrent bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cephalexin; Anti-Bacterial Agents; Surgical Procedures, Operative; Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cipro (Experimental): ciprofloxacin
  Interventions: Procedure: surgical procedure; Drug: Ciprofloxacin
- ceph (Experimental): cephalexin
  Interventions: Drug: cephalexin; Procedure: surgical procedure

INTERVENTIONS:
Drug: cephalexin — 500 mg oral bid for 3 days starting the night before resection
  Other Names: antibiotic
  Arms: ceph
Procedure: surgical procedure
Drug: Ciprofloxacin — 500 mg oral bid for 3 days starting the night before resection
  Other Names: cipro
  Arms: cipro

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. It is not yet known whether ciprofloxacin is more effective than cephalexin in preventing cancer recurrence in patients who are undergoing surgery to treat bladder cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of ciprofloxacin with that of cephalexin in preventing recurrence of cancer in patients who are undergoing surgery for bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether ciprofloxacin improves the recurrence-free survival of patients with superficial transitional cell carcinoma of the bladder treated with a transurethral tumor resection.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to disease status (first occurrence vs recurrent disease). Patients are randomized to receive either oral ciprofloxacin or oral cephalexin 2 times a day for 3 days starting the night before resection. Patients who are allergic to penicillin or a cephalosporin receive oral co-trimoxazole 2 times a day for 3 days. All patients undergo complete resection of all bladder tumors. Patients are followed every 3 months for the first 2 years, every 6 months for the next 2 years, and at the end of the fifth year.

PROJECTED ACCRUAL: A total of 900 patients will be accrued for this study over 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Stage Ta (any grade) transitional cell carcinoma of the bladder on basis of cystoscopy Recurrent disease no greater than T1 Must not be at high risk for upper tract (ureter or renal pelvic) transitional cell cancers

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: SWOG 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Not pregnant or nursing Fertile patients must use effective contraception No other prior malignancy in the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer in complete remission No allergies to fluoroquinolones If allergic to penicillin or cephalosporin, must be able to take co-trimoxazole

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 28 days since prior intravesical therapy and recovered Endocrine therapy: Not specified Radiotherapy: At least 28 days since prior radiotherapy and recovered Surgery: Not specified Other: At least 3 months prior to cystoscopy since prior fluoroquinolones No concurrent fluoroquinolones No concurrent hemodialysis or peritoneal dialysis No concurrent probenecid or theophylline No concurrent antacids containing aluminum, magnesium or calcium, products containing iron or zinc, caffeine, cyclosporine, or warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 1999-04; Primary Completion 2001-07 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P. Wood, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (90):
- United States (90):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - Eastern Virginia Medical School, Norfolk, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington

REFERENCES:
- [Result] Wolman SR, Goldman B, Slovak ML, Tangen C, Persons DL, Wood D. Aneusomy for detection of bladder cancer recurrence: a Southwest Oncology Group study. Cancer Genet Cytogenet. 2007 Jul 1;176(1):22-7. doi: 10.1016/j.cancergencyto.2007.02.015. PMID 17574960